CLINICAL TRIAL: NCT06731621
Title: Psilocybin for Treatment-Resistant Depression in Autism: a Pilot Trial With Pre-Post Brain and Cognitive Measurement to Understand Mechanism
Brief Title: Psilocybin for Treatment-Resistant Depression in Autism
Acronym: PAT-DA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/112
Record Dates: First submitted 2024-11-19; First posted 2024-12-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-01

CONDITIONS: Treatment Resistant Depression; Autism Spectrum Disorder
Keywords: Treatment Resistant Depression; Autism Spectrum Disorder; psilocybin-assisted therapy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Autism Spectrum Disorder | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label (Experimental): Safety Dosing Session (V3): 10mg of psilocybin + therapy + safety evaluations
  Active Treatment Session (V4): 25mg of psilocybin + therapy + safety evaluations
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 2 dosing sessions 1 week apart, each about 6-8 hours duration
  Psilocybin-assisted therapy (PAT), is a psychotherapeutic intervention in which the psychological effects of psilocybin play a significant role. PAT procedures typically involve psychological preparation prior to therapist-supported psilocybin dosing sessions. These sessions are used to establish a therapeutic relationship, inform participants about what to expect, and set expectations for the dosing session. During the psilocybin dosing session, trained therapists support the individual through their experience and psychological integration therapy occurs after the dosing experience. PAT has shown impressive antidepressant effects in people with TRD or severe MDD in at least six modern-era clinical trials (Andersen et al., 2021).
  Other Names: Psilocybin-Assisted Therapy

SUMMARY:
We propose a first-of-its-kind open-label clinical trial to investigate the feasibility, tolerability, and safety of administering psilocybin in autistic adults with treatment-resistant depression (TRD). In this study, 20 participants (intellectually able and fluent-speech adults) with autism and co-occurring TRD will receive around 20 hours of manualized psychotherapy that has previously been used with psilocybin (Agin-Liebes et al., 2020). They will also receive psilocybin at 2 different time points, firstly a safety dose of 10mg, followed by a treatment dose of 25mg. This study design is in accordance with previous studies investigating the use of psilocybin with psilocybin-assisted therapy (PAT) to treat TRD (Carhart-Harris et al., 2016, 2018)

DETAILED DESCRIPTION:
Each participant will begin with a screening visit (V1), during which eligibility will be determined through clinical and psychiatric assessments of the participant's physical and mental health. Following confirmation of eligibility, the study procedures will begin.

The participant will begin with a 2-4 week tapering period during which they will taper and discontinue any conventional antidepressants. Most conventional antidepressants will require a minimum 2-week tapering period, with the exception of fluoxetine, which will require a 4-week tapering period. Additional time may be added at the discretion of the study investigator. During the tapering period, there will be weekly check-ins with a study psychiatrist by in-person assessment or brief telephone calls to monitor for worsening depression and suicidality. Following the tapering period, participant eligibility will be re-assessed for the eligibility.

At Study Visit 2 (Baseline, V2), participants will complete a series of questionnaires and assessments (Table 2) and preparatory therapy with trained study therapists. The participant will also receive a brain MRI scan lasting for about 45 minutes.

At Study Visits 3 & 4 (V3/V4), participants will receive oral doses of psilocybin (safety dose of 10 mg at V3, treatment dose of 25 mg at V4), to assess the tolerability and efficacy of psilocybin. These sessions will be held one week apart and will last 6 to 8 hours each. These sessions will take place in a pre-decorated treatment room at CAMH. Throughout the entire duration of the dosing sessions, participants will be monitored by a minimum of two trained therapists. At the end of each session, participants will be evaluated for safety by a study psychiatrist before being discharged. Participants will also rate the 11-Dimension Altered States of Consciousness (11D-ASC) at the end of each dosing day when the subjective effects of psilocybin have subsided to a negligible level. In addition, the participant will also receive a second brain MRI scan lasting for about 30 minutes (V3a) following V3 Safety dosing. To reduce participant burden, MRI scan can be completed on the following day or within 1-3 days following safety dosing (V3). The participants will also be required to complete the self-rated questionnaires at this additional MRI assessment.

Visit 5 (V5) will be held one day after administration of the treatment dose (V4). During V5 the participants will complete post-treatment clinical and cognitive assessments, alongside the third and final MRI scan (of the main clinical trial design). Participants will also undergo a 1-hour integration therapy session to debrief their experiences the day before. Visit 6 (V6) will be held one week following the treatment dose (V4). During V6 a second 1-hour integration therapy session takes place and all post-treatment clinical assessments will be repeated. Subsequent clinical progress will be evaluated virtually at V7, V8, V9, which will respectively be held 2, 4, and 12 weeks following the treatment session (V4).

10 participants out of 20 participants in the main clinical trial could opt to receive 7 additional brain MRI scans besides the MRI scans at V2, V3a and V5 required in the main clinical trial. These 7 additional scans will be assessed at V1, in the middle of medication washout/tapering period V6, V7, V8, 8 weeks following the treatment dose (V4), and V9, respectively. At each optional MRI visit, self-rated assessments will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Must be aged 18 to 65 years old;
2. Must be deemed to have capacity to provide informed consent;
3. Ability to read and communicate in English;
4. Must sign and date the informed consent form;
5. Stated willingness to comply with all study procedures;
6. Intellectually able: Either 1) the participant has a previous report showing intelligence quotient (IQ) ≥ 70 on the General Abilities Index of the Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) or any other standardized intelligence scales, or 2) the participant scores >10 percentile on the nine-item form of the Raven's Standard Progressive Matrices Test (RSPM).
7. Clinical diagnosis of autism spectrum disorder (ASD), based on the DSM-5 or ICD-11
8. Primary DSM-5 diagnosis of non-psychotic MDD, single or recurrent, based on the Mini International Neuropsychiatric Interview (MINI) administered at the first screening visit (V1);
9. Participants diagnosed with treatment-resistant depression defined as individuals with a baseline GRID-HAMD-17 score > 14 and that have not responded to two or more separate trials of antidepressants at an adequate dosage and duration based on the Antidepressant Treatment History Form; there is no upper limit on the number of treatment failures;
10. Ability to take oral medication;
11. Individuals who are capable of becoming pregnant: use of highly effective contraception for at least 3 months prior to screening and agreement to use such a method during study participation;
12. Individuals who are willing to taper off current antidepressant and antipsychotic medications for a minimum of 2-weeks (or more depending on the medication) prior to Baseline (V2) and whose physician confirms that it is safe for them to do so; and
13. A clean urine drug screen and negative urine pregnancy test (in females).
14. Agreement to adhere to Lifestyle Considerations (see below) throughout study duration

Exclusion Criteria:

1. Pregnant as assessed by a urine pregnancy test or individual's that intend to become pregnant during the study or are breastfeeding;
2. Treatment with another investigational drug or other intervention within 30 days of Screening (V1);
3. The presence of an unstable seizure disorder as defined by having not been seizure-free for at least 6 months or anticonvulsant treatment has not been stable for at least 4 weeks;
4. The presence of any clinically significant or unstable medical conditions, including cardiovascular, liver, kidney, pulmonary disease, presence of known congenital brain malformation, as per investigator assessment based on medical history and chart review;
5. Moderate or severe DSM-5 diagnosis of an alcohol or substance use disorder in the past 12 months;
6. Any DSM-5 lifetime diagnosis of a schizophrenia-spectrum disorder, psychotic disorder (unless substance induced or due to a medical condition), bipolar I or II disorder, paranoid personality disorder, or neurocognitive disorder as determined by medical history and the MINI clinical interview;
7. Any first-degree relative with a diagnosis of schizophrenia-spectrum disorder; psychotic disorder (unless substance-induced or due to a medical condition); or bipolar I or II disorder as determined by the family medical history form and discussions with the participant;
8. Presence of a relative or absolute contraindication to psilocybin, including a drug allergy, recent stroke history, uncontrolled hypertension, low or labile blood pressure, recent myocardial infarction, cardiac arrhythmic, severe coronary artery disease, or moderate to severe renal or hepatic impairment;
9. Substantial lifetime use (>10 years total) or recent use (past 6 months) of ketamine, psychedelics, or MDMA and positive urine toxicological screen at Screening (V1) and Baseline (V2);
10. Any other clinically significant physical illness, including chronic infectious diseases or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if they take part in the study;
11. Have active suicidal ideation with intent and plan as determined by SBQ-ASC.
12. Have initiated new psychotherapy within 12 weeks prior to Screening
13. Contraindication to MR imaging or a previous history of claustrophobia.

Lifestyle considerations:

During this clinical trial, participants are asked to:

* Abstain from alcohol for 24 hours before the intervention or the day of the intervention (V3, V4).
* Abstain from the use of any prescribed opioids, benzodiazepines, or sleep aids (Z-drugs) within 12 hrs prior to the intervention (V3, V4) and for up to 6 hrs after administration.
* Abstain from any illicit drugs (e.g. cocaine, ecstasy/MDMA, hallucinogens) for the duration of the study.
* Abstain from any cannabinoids within 3 weeks prior to the intervention (V3, V4) and until the completion of the 2nd integrative therapy session (V6).
* Abstain from driving or operating heavy machinery for up to 24 hours after the intervention (V3, V4).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Administering Psilocybin in Conjunction with Psychotherapy in Autistic Adults | From enrollment to end of treatment & follow-up at 12 weeks post-intervention (12 weeks post treatment dosing i.e., Day 0)
  Percentage of participants recruited and retained.
Subjective Psychedelic Effects as Measured by the 11-Dimensions of Altered States of Consciousness (11D-ASC) Rating Scale | Administered following each dosing session (Visit 3 (Safety dosing - Day -7)) & Visit 4 (treatment dosing - Day 0))
  A visual analogue scale (0-100 millimeters in length) with higher scores indicating more intense effects. Each question is attributable to one of the specified 11 dimensions of altered states of consciousness.
Number of Participants with Treatment-Related Adverse Events as Assessed by SBQ-ASC & UKU Side Effect Rating Scale | From enrollment to end of treatment & follow-up at 12 weeks post-intervention (12 weeks post treatment dosing i.e., Day 0)
  Treatment-Related Adverse Events are expected to be similar in nature & frequency to those reported in previous clinical studies on classic psychedelics in neurotypical populations.
  The UKU Side Effect Scale will be used to capture & document core features of any treatment-related side effects. The Suicidal Behaviors Questionnaire - Autism Spectrum Conditions (SBQ-ASC) will be used to measure suicidality in participants. It consists of 5 scored items: 1) lifetime experience of suicidal thoughts; 2) frequency of intense suicidal thoughts in the last 12 months; 3) perseverative intense suicidal thoughts; 4) likelihood of suicide attempts; 5) communication of future suicide intent & past suicide attempts to others. The SBQ-ASC also includes optional follow-up items which are not scored, based on responses to Item 5: for those who have attempted suicide, the follow-up items address presence of plans, impulsivity, and access to means.
Feasibility of Dense Sampling Brain MRI Procedures & Trial Design | From enrollment to end of treatment & follow-up at 12 weeks post-intervention (12 weeks post-treatment dosing i.e., Day 0)
  Percentage of participants recruited and retained for the optional dense sampling brain MRI procedures (multiple scans throughout duration of participant's involvement in study, up to 10 ).

SECONDARY OUTCOMES:
Changes in Brain Network Interactions as Assessed with Pre- and Post-Intervention MRI Brain Scans | Evaluated using MRI before and after each dosing session (Visit 2 (Baseline Visit - Day -15 to -8)), Visit 3a (one day after safety dosing - Day -6)) & Visit 5 (one day after treatment dosing - Day 1))
  Brain MRI scans and subsequent brain network & cognitive modelling will be used to assess & study changes in brain network interactions and possible mechanisms underpinning antidepressant effects of psilocybin for treatment-resistant depression in autism.
Changes & Variance in Brain Functional Connectivity Assessed Across Dense Sampling Brain MRI Sessions | From enrollment to end of treatment & follow-up at 12 weeks post-intervention (12 weeks post treatment dosing i.e., Day 0)
  The optional dense sampling brain MRI procedures will allow for a more robust model of the brain and changes/variance that may be observed in an individual's brain over the course of the study, particularly in response to the intervention. Brain MRI scans and subsequent brain network & cognitive modelling will be used to assess & study changes in brain network interactions and possible mechanisms underpinning antidepressant effects of psilocybin for treatment-resistant depression in autism.

OTHER OUTCOMES:
Antidepressant Efficacy of Psilocybin-Assisted Psychotherapy for Autistic Adults with Treatment-Resistant Depression | From enrollment to end of treatment & follow-up at 12 weeks post-intervention
  The following measures will assess antidepressant efficacy:
  Clinical Global Impression Scale (CGI) - Clinician-administered scale providing a brief, stand-alone assessment of the clinician's view of the participant's global functioning before and after initiating study medication. 7-point scale; higher scores indicate more severe symptoms.
  Beck Depression Inventory II (BDI-II) - 4-point scale measuring severity of depression and related symptoms; higher scores indicate more severe depressive symptoms.
  Snaith-Hamilton Pleasure Scale (SHAPS) - 4-point scale measuring hedonic capacity; lower scores indicate greater hedonic capacity (less anhedonia).
  Ruminative Responses Scale (RRS-10) - 4-point scale describing responses to depressed mood; higher scores reflect more severe rumination.
  Anxiety Scale for Autism - Adults (ASA-A) - 4-point scale measuring anxiety in autistic adults; higher scores indicate greater anxiety.
Changes in Psychological Symptoms & Features Theoretically Associated with Psilocybin-Assisted Psychotherapy & Depression | Administered at follow-up visits post-intervention (Visits 5-9)
  General Alexithymia Factor Score (GAFS-8) - Self-report assessing difficulty identifying and describing feelings.
  Acceptance & Action Questionnaire-II (AAQ-II) - Self-report measuring experiential avoidance and psychological inflexibility.
  Autism Burnout Survey Items (ABSI) - Self-report quantifying autistic burnout (exhaustion, withdrawal, cognitive overload) from stressors amplified in autistic individuals.
  Connor-Davidson Resilience Scale 10 (CD-RISC-10) - Measures resilience and flexibility in adapting to stressful situations.
  Interoception Sensory Questionnaire-8 (ISQ-8) - Measures perception and interpretation of interoceptive capacity.
  Interpersonal Needs Questionnaire (INQ-15) - Assesses 'thwarted belongingness' and 'perceived burdensomeness'.
  Cognitive Flexibility Inventory (CFI) - Self-report assessing cognitive flexibility in challenging and replacing maladaptive thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yuan Lin, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
In the publication of the results of research, the investigators are obliged to preserve the confidentiality of all research participants. Participants will not be identified in any publication of research results. The results of this study will be published as group data without the use of characteristics that would identify individual participants. The study investigator will hold the primary responsibility for the publication of the results of the clinical trial. All publications will follow CAMH policies associated with publications.